CLINICAL TRIAL: NCT02200783
Title: Randomized Comparison of Radiological Exposure Between Radial and Femoral Technique Assessing Use of Protective Device Dedicated TRIPTable® in Patients With Acute Coronary Syndromes Undergoing Cardiac Catheterization
Brief Title: Randomized Comparison of Radiological Exposure With TRIPTable® in Patients With Acute Coronary Syndromes
Acronym: TRIPTABLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Marilia Medicine School (Other)
Responsible Party: Principal Investigator, Igor Bienert, MD, Marilia Medicine School
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 718016; CAAE 32767514.0.0000.5413 (Other: Plataforna Brasil)
Record Dates: First submitted 2014-07-23; First posted 2014-07-25 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Acute Coronary Syndromes; Angioplasty, Transluminal, Percutaneous Coronary
Keywords: Cardiac catheterization; Radiation Protection; Radial artery; Femoral artery
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Keratotomy, Radial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Radial (Active Comparator): Cardiac catheterization and coronary angioplasty performed via standard radial artery technique.
  Interventions: Device: Radial
- Femoral (Active Comparator): Cardiac catheterization and coronary angioplasty performed via standard femoral artery technique.
  Interventions: Device: Femoral
- TripTable (Experimental): Cardiac catheterization and coronary angioplasty performed with standard transradial technique plus using the TRIPTable device.
  Interventions: Device: TripTable

INTERVENTIONS:
Device: TripTable — Details of the device previously described, designed to medical operator radioprotection. No changes in radial technique beyond the use of the supportive device will be performed.
  Other Names: TRansradial Intervention Protection Table
  Arms: TripTable
Device: Radial — Standard radial artery catheterization procedure, performed for the purpose of coronary angiography and ad hoc angioplasty if necessary.
  Other Names: PHILIPS standard cath arm support - NCVA097
  Arms: Radial
Device: Femoral — Standard femoral artery catheterization procedure, performed for the purpose of coronary angiography and ad hoc angioplasty if necessary. The supporting device will be the patient's own body, placing the material above the legs.
  Arms: Femoral

SUMMARY:
Excessive radiation received by the operator has been described as a possible drawback of the radial catheterization technique when compared with the femoral access.

The study hypothesis is that the use of radial access device dedicated radioprotective TRIPTable ® (Transradial Intervention Table Protection) is not inferior to standard femoral technique and superior to standard radial technique as radioprotection strategy to the operator in patients with acute coronary syndromes acute and submitted to cardiac catheterization.

DETAILED DESCRIPTION:
This study is prospective, 1:1:1 randomized, unicentric, comparative between femoral and radial radial technique with and without dedicated TRIPTable ® device.

The TripTable device is a polycarbonate support table anatomically-designed to facilitate the radial technique, facilitating the puncturing, positioning, support to work material and providing further radioprotection from a lead layer without obstruction in viewing the fluoroscopic images.

ELIGIBILITY:
Inclusion Criteria:

* Unstable angina with an indication for invasive stratification
* Acute coronary syndrome without ST-segment elevation
* Acute coronary syndrome with ST-segment elevation
* Patient informed of the nature of the study and have signed the Informed Consent
* Patient suitable for coronary angiography and / or percutaneous coronary intervention either by radial access as the femoral

Exclusion Criteria:

* Below 18 years of age
* Pregnancy
* Chronic use of vitamin K antagonists, or direct thrombin inhibitors or antagonists of factor Xa,
* Active bleeding or high risk of bleeding (severe hepatic insufficiency, active peptic ulcer disease, creatinine clearance <30 mL / min, platelet count <100,000 mm3);
* Uncontrolled hypertension;
* Cardiogenic shock;
* Previous coronary artery bypass graft surgery with the use of ≥ 1 graft
* Patients not candidates for the use of any of the specified vascular access
* Concomitant severe disease with life expectancy less than 12 months life;
* Medical, geographical, or social conditions that impede study participation
* Refusal or inability to understand and sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Radiation dose | 1 year
  Accumulated radiation dose received by the operator during the interventional cardiology procedures as measured by Thermoluminescent Dosimeters (TLD)

SECONDARY OUTCOMES:
Radiation according measured site | 1 year
  accumulated radiation dose received by each measured site (gonadal, thyroid and lens)
Operator absorbed radiation according total radiation dose | 1 year
  Evaluation of radiation dose to the operator according to linear correlation corrected for total dose of radiation.
Success of procedure | 1 year
  Success rate of the procedure, as defined by perform the procedure without need to cross between techniques

OTHER OUTCOMES:
Clinical data | 1 year
  Registration of clinical features and procedural data, to compare with historical control group (ARISE trial - NCT01653587) using similar inclusion criteria without the objectives of the current study operator (to exclude Hawthorne effect).

CONTACTS AND LOCATIONS:
Overall Officials: Igor RC Bienert, MD, Study Director — Marilia School of Medicine
Locations (1):
- Marilia School of Medicine, Marília, São Paulo, Brazil

REFERENCES:
- [Background] Chambers CE, Fetterly KA, Holzer R, Lin PJ, Blankenship JC, Balter S, Laskey WK. Radiation safety program for the cardiac catheterization laboratory. Catheter Cardiovasc Interv. 2011 Mar 1;77(4):546-56. doi: 10.1002/ccd.22867. Epub 2011 Jan 19. PMID 21254324
- [Background] Sciahbasi A, Romagnoli E, Trani C, Burzotta F, Sarandrea A, Summaria F, Patrizi R, Rao S, Lioy E. Operator radiation exposure during percutaneous coronary procedures through the left or right radial approach: the TALENT dosimetric substudy. Circ Cardiovasc Interv. 2011 Jun;4(3):226-31. doi: 10.1161/CIRCINTERVENTIONS.111.961185. Epub 2011 May 17. PMID 21586692
- [Background] Sciahbasi A, Calabro P, Sarandrea A, Rigattieri S, Tomassini F, Sardella G, Zavalloni D, Cortese B, Limbruno U, Tebaldi M, Gagnor A, Rubartelli P, Zingarelli A, Valgimigli M. Randomized comparison of operator radiation exposure comparing transradial and transfemoral approach for percutaneous coronary procedures: rationale and design of the minimizing adverse haemorrhagic events by TRansradial access site and systemic implementation of angioX - RAdiation Dose study (RAD-MATRIX). Cardiovasc Revasc Med. 2014 Jun;15(4):209-13. doi: 10.1016/j.carrev.2014.03.010. Epub 2014 Mar 26. PMID 24746599
- [Background] Park EY, Shroff AR, Crisco LV, Vidovich MI. A review of radiation exposures associated with radial cardiac catheterisation. EuroIntervention. 2013 Oct;9(6):745-53. doi: 10.4244/EIJV9I6A119. PMID 24169135
- [Result] de Andrade PB, E Mattos LA, Tebet MA, Rinaldi FS, Esteves VC, Nogueira EF, Franca JI, de Andrade MV, Barbosa RA, Labrunie A, Abizaid AA, Sousa AG. Design and rationale of the AngioSeal versus the Radial approach In acute coronary SyndromE (ARISE) trial: a randomized comparison of a vascular closure device versus the radial approach to prevent vascular access site complications in non-ST-segment elevation acute coronary syndrome patients. Trials. 2013 Dec 18;14:435. doi: 10.1186/1745-6215-14-435. PMID 24345099
- [Result] Jolly SS, Yusuf S, Cairns J, Niemela K, Xavier D, Widimsky P, Budaj A, Niemela M, Valentin V, Lewis BS, Avezum A, Steg PG, Rao SV, Gao P, Afzal R, Joyner CD, Chrolavicius S, Mehta SR; RIVAL trial group. Radial versus femoral access for coronary angiography and intervention in patients with acute coronary syndromes (RIVAL): a randomised, parallel group, multicentre trial. Lancet. 2011 Apr 23;377(9775):1409-20. doi: 10.1016/S0140-6736(11)60404-2. Epub 2011 Apr 4. PMID 21470671
- [Result] Romagnoli E, Biondi-Zoccai G, Sciahbasi A, Politi L, Rigattieri S, Pendenza G, Summaria F, Patrizi R, Borghi A, Di Russo C, Moretti C, Agostoni P, Loschiavo P, Lioy E, Sheiban I, Sangiorgi G. Radial versus femoral randomized investigation in ST-segment elevation acute coronary syndrome: the RIFLE-STEACS (Radial Versus Femoral Randomized Investigation in ST-Elevation Acute Coronary Syndrome) study. J Am Coll Cardiol. 2012 Dec 18;60(24):2481-9. doi: 10.1016/j.jacc.2012.06.017. Epub 2012 Aug 1. PMID 22858390